CLINICAL TRIAL: NCT02327442
Title: Prospective Imaging Study of 68Ga-NOTA-NFB in Tumors
Brief Title: 68Ga-NOTA-NFB: Radiation Dosimetry in Healthy Volunteers and Applications in Glioma Patients or Breast Cancer Patients
Acronym: GNNGB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20140522-6
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Glioma; Breast Cancer
Keywords: chemokine receptor; galium; dosimetry; glioma
MeSH Terms: conditions — Glioma; Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Volunteers: Healthy Volunteers undergo whole-body 68Ga-NOTA-NFB PET/CT scans 0, 0.5, 1.0, 2.0, and 3.0 hours after tracer injection. During the imaging period, 1 mL blood samples are obtained specifically at 1, 3, 5, 10, 30,60, 90, 120, 150, and 180 minutes after the injection, for time-activity curve calculations.
  Interventions: Radiation: 68Ga-NOTA-NFB
- Glioma Patients: Glioma Patients enrolled for the clinical study of diagnosing glioma are performed with both 68Ga-NOTA-NFB PET/CT and18F-FDG PET/CT scans before surgery.
  Interventions: Radiation: 68Ga-NOTA-NFB
- Breast Cancer Patients: 68Ga-NOTA-NFB PET/CT and 18F-FDG PET/CT scans will undergo in patients with breast cancer before and after neoadjuvant chemotherapy.
  Interventions: Radiation: 68Ga-NOTA-NFB

INTERVENTIONS:
Radiation: 68Ga-NOTA-NFB — In this investigation, 68Ga-NOTA-NFB is employed to a preclinical trial, including radiation dosimetry study in healthy volunteers and the first application in glioma patients, to assess the safety, dosimetry property and evaluate the CXCR4 expression in glioma patients and breast cancer patients.

SUMMARY:
The purpose of this study is to assess the safety, biodistribution, dosimetric properties of the positron emission tomography (PET) radiopharmaceutical agent 68Ga-NOTA-NFB. To preliminarily evaluate its application in glioma diagnosis.

To assess the application of 68Ga-NOTA-NFB PET/CT in the evaluation of the neoadjuvant chemotherapy in patients with breast cancer before and after the therapy.

DETAILED DESCRIPTION:
6 healthy volunteers with whole-body PET/CT scans 0, 0.5, 1.0, 2.0, and 3.0 hours after tracer injection (mean dose, 4.93 ± 0.10 mCi) will be performed. During the imaging period, 1 mL blood samples will be obtained specifically at 1, 3, 5, 10, 30,60, 90, 120, 150, and 180 minutes after the injection, for time-activity curve calculations. The estimated radiation doses will be calculated by using OLINDA/EXM software.

8-10 patients with glioma will be enrolled for the clinical study of diagnosing glioma, they will be performed with both 68Ga-NOTA-NFB PET/CT and18F-FDG PET/CT scans before surgery. The preoperative images are compared and correlated with the pathologically report. Next, the expression of CXCR4 will be determined by immunohistochemical staining of the resected brain tumor tissues.

30 patients with breast cancer will be underwent 68Ga-NOTA-NFB PET/CT and18F-FDG PET/CT scans before and after the neoadjuvant chemotherapy. SUV of lesions before and after therapy will be contrasted.

ELIGIBILITY:
Inclusion Criteria:

* volunteers : healthy patients with glioma: diagnosed by MR and ready for surgery patients with breast: cancer appropritate of neoadjuvant chemotherapy.

Exclusion Criteria:

* patients with glioma: refuse or cannot endure surgery. patients with breast: refuse neoadjuvant chemotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 6 healthy volunteers. 10 patients with glioma before surgery. 30 patients with breast cancer before and after neoadjuvant chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
SUV of organs | 0, 0.5, 1.0, 2.0, and 3.0hours after injection
  The standardized uptake values (SUV) in deferent organs are calculated.
radioactivity of blood sample | 1, 3, 5, 10, 30,60, 90, 120, 150, and 180minutes
  blood samples are obtained specifically at 1, 3, 5, 10, 30,60, 90, 120, 150, and 180 minutes after the injection, for time-radioactivity curve calculations.
SUV of glioma | 1 hour after injection
  The maximum standardized uptake values (SUVmax) and the maximum target to non-target ratios (T/NTmax) of 68Ga-NOTA-NFB and 18F-FDG in glioma tissues.
SUV of Breast Cancer | 1 hour after injection
  The maximum standardized uptake values (SUVmax) of 68Ga-NOTA-NFB and 18F-FDG in breast cancer before and after neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, Doctor, Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital Nuclear Medicine Department, Xi'an, Shaanxi, China